CLINICAL TRIAL: NCT02765815
Title: A Prospective Randomized Case Series Comparison on the Clinical Efficacy of Exparel Local Anesthetic in Total Knee Arthroplasty Patients
Brief Title: A Comparison of Exparel Local Anesthetic in Total Knee Arthroplasty (TKA) Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: competing protocol
Sponsor: Holy Cross Hospital, Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Exparel TKA
Record Dates: First submitted 2016-01-27; First posted 2016-05-09 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis, Knee; Arthroplasty, Replacement, Knee
Keywords: TKA; Knee replacement; Arthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis | interventions — Bupivacaine; Epinephrine; Ketorolac; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel plus multi-drug cocktail (Active Comparator): Liposomal bupivacaine, 266mg plus Bupivacaine 0.25% with Epinephrine, Ketorolac 30mg, and Morphine 10mg.
  Interventions: Drug: Liposomal bupivacaine, 266mg; Drug: Ketorolac 30mg; Drug: Morphine 10mg; Drug: Bupivacaine 0.25% with Epinephrine
- Multi-drug cocktail alone (Active Comparator): Bupivacaine 0.5% with Epinephrine, Ketorolac 30mg, Morphine 10mg.
  Interventions: Drug: Bupivacaine 0.5 % with Epinephrine; Drug: Ketorolac 30mg; Drug: Morphine 10mg

INTERVENTIONS:
Drug: Liposomal bupivacaine, 266mg
  Other Names: Exparel Injection
  Arms: Exparel plus multi-drug cocktail
Drug: Bupivacaine 0.5 % with Epinephrine
  Arms: Multi-drug cocktail alone
Drug: Ketorolac 30mg
Drug: Morphine 10mg
Drug: Bupivacaine 0.25% with Epinephrine
  Arms: Exparel plus multi-drug cocktail

SUMMARY:
This is a prospective, single-center, single-blinded, randomized, case-control study. The study is conducted by a single investigator at an orthopedic surgery institute, with a minimum 6 week post operative follow-up period of TKA patients who receive Exparel compared with the surgeon's standard method (detailed below) for pain management intraoperatively.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-blinded, randomized, case-control study. The study is conducted by a single investigator at an orthopedic surgery institute, with a minimum 6 week post operative follow-up period. Subjects scheduled for a planned total knee arthroplasty procedure will be consented and those meeting study criteria will be randomized to receive intra-operative injections at the surgical site of liposomal bupivicaine plus a multi-drug cocktail, or a multi-drug cocktail alone.

This study will recruit subjects on an ongoing basis with a minimum of 130 study participants and a maximum of 156. Efficacy data on surgical pain control and safety data will be collected at frequent intervals during the hospitalization. Each study participant will be followed for a minimum 6 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 88 years of age.
2. Subject is scheduled to undergo primary unilateral Total Knee Arthroplasty.
3. Subject willing and able to sign the informed consent.
4. Subject is fluent in verbal and written English.
5. Subject agrees to take Liposomal bupivacaine or standard of care equivalent.

Exclusion Criteria:

1. Previous Partial or Total Knee Arthroplasty of the study knee. Previous Non-Implant surgery on the study knee and contralateral knee is permitted.
2. Subject is pregnant or planning to become pregnant while enrolled in the study.
3. Subject has a history of narcotic or alcohol abuse.
4. Subjects with hepatic disease or renal impairment (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x upper limit of normal or estimated glomerular filtration rate (eGFR) < 30 ml/min within 30 days of surgery).
5. For any reason, in the opinion of the investigator, the Subject may not be a suitable candidate for study participation (i.e., history of noncompliance, drug dependency, etc.)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Estimated); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Patient reported Visual Analog Scale (VAS) pain intensity score. Post-surgery hours 4-24. | VAS pain intensity scores will be collected starting four hours after end of surgery and every 4 hours thereafter until hour 24.
  The area under the curve (AUC) of the VAS scores from 4-24 hours will be compared between the two treatment groups.
Patient reported VAS pain intensity score. Post-surgery hours 24-48. | VAS pain intensity scores will be collected starting 24 hours after end of surgery and every 4 hours thereafter until hour 48, or discharge.
  The AUC of the VAS scores from 24-48 hours or until discharge will be compared between the two treatment groups.
Patient reported VAS pain intensity score. Post-surgery hours 48-72. | VAS pain intensity scores will be collected starting 48 hours after end of surgery and every 4 hours thereafter until hour 72, or discharge.
  The AUC of the VAS scores from 48-72 hours or until discharge will be compared between the two treatment groups.

SECONDARY OUTCOMES:
Cost:benefit analysis | TKA hospitalization charges, and VAS pain intensity scores pre-operative on day of surgery, 2-week and 6-week followup visits.
  Correlation between hospital charges and improvement in VAS pain intensity score from baseline to the 2-week and 6-week follow-up time points.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Roche, MD, Principal Investigator — Holy Cross Orthopedic Research Institute
Locations (1):
- Holy Cross Hospital Orthopedic Research Institute, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Result] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Result] Fetherston CM, Ward S. Relationships between post operative pain management and short term functional mobility in total knee arthroplasty patients with a femoral nerve catheter: a preliminary study. J Orthop Surg Res. 2011 Feb 7;6:7. doi: 10.1186/1749-799X-6-7. PMID 21294923
- [Result] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Result] Bagsby DT, Ireland PH, Meneghini RM. Liposomal bupivacaine versus traditional periarticular injection for pain control after total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1687-90. doi: 10.1016/j.arth.2014.03.034. Epub 2014 Apr 4. PMID 24793570
- [Result] Broome CB, Burnikel B. Novel strategies to improve early outcomes following total knee arthroplasty: a case control study of intra articular injection versus femoral nerve block. Int Orthop. 2014 Oct;38(10):2087-9. doi: 10.1007/s00264-014-2392-0. Epub 2014 Jun 18. PMID 24938586
- [Result] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545